CLINICAL TRIAL: NCT00553449
Title: A Randomised, Controlled, Parallel-group, Open-label Study to Evaluate Different Dosing Regimens of Rabeprazole in Controlling Nocturnal Heartburn Symptoms in Patients With Gastroesophageal Reflux Disease.
Brief Title: Open Label Study Evaluating Different Dosing Regimens of Rabeprazole in Gastro-esophageal Reflux Disease (GERD) Patients With Night-time Heartburn Symptoms.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005692
Record Dates: First submitted 2007-11-01; First posted 2007-11-05 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-03

CONDITIONS: Gastroesophageal Reflux; Heartburn
Keywords: nocturnal heartburn; day-time heartburn; rabeprazole; GERD
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Rabeprazole

INTERVENTIONS:
Drug: rabeprazole

SUMMARY:
The purpose of this study is to evaluate the effect of each of the rabeprazole treatment regimens on nocturnal heartburn symptoms.

DETAILED DESCRIPTION:
There is limited data regarding the estimate of patients who experience nocturnal symptoms despite adequate daytime heartburn control, the incidence and severity of nocturnal heartburn episodes after a minimum of 4 weeks of acid suppressive therapy with a Proton-pump inhibitor (PPI) or Histamine -2-receptor antagonist (H2RA), and the effect of instituting rabeprazole therapy after failure to control nocturnal heartburn symptoms with other acid suppressive therapy. This is a multicentre, randomised (study medication is assigned by chance), controlled, parallel-group, open-label study in GERD patients. Patients will be screened and enter a 2-week run-in phase to document heartburn symptoms while on their current therapy, during which they will complete a daily diary of symptoms and antacid use. Patients who have troublesome nocturnal heartburn episodes, but adequate daytime heartburn symptom control (as defined) will enter an 8-week treatment phase where they are randomised to one of the rabeprazole regimens: 20mg once daily in the evening (dose administered 30minutes prior to the evening meal; "QPM" regimen), 10mg twice daily (dose administered 30minutes prior to the morning and evening meals; "BID/twice daily" regimen) or 20mg once daily in the morning (dose administered 30minutes prior to the morning meal; "QAM/every morning" regimen), plus antacids as required. The study hypothesis is that after failure to control night-time heartburn symptoms with other acid suppressive therapy, instituting rabeprazole will have a beneficial effect. Safety assessments include: physical examination and pregnancy test at screening, vital signs and weight at randomization and final visit, adverse event and concomitant medication reporting at every visit. Rabeprazole 20mg once daily in the evening: one rabeprazole 20mg tablet daily in the evening, 30-60 minutes before dinner for 56 days OR Rabeprazole 10mg twice daily: one rabeprazole 10mg tablet in the morning, 30-60 minutes before breakfast, and one rabeprazole 10mg tablet 30-60 minutes before dinner for 56 days. OR Rabeprazole 20mg once daily in the morning: one rabeprazole 20mg tablet daily in the morning, 30-60 minutes before breakfast for 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had a minimum three-month history of symptomatic GERD, with heartburn as the predominant symptom, and must report nocturnal heartburn symptoms (i.e., heartburn symptoms experienced during the night-time period, between 2200 and 0600h)
* Patients must currently be taking a proton-pump inhibitor (PPI) or histamine-2 receptor antagonist (H2RA) at least four weeks prior to study admission
* Patients must be able to read, write and understand the language of the HRQOL and productivity assessment instruments (PAGI-SYM, PAGI-QOL, WPAI-GH) i.e., English or French
* Patients must have been at least 80% compliant with their current acid suppressive therapy, and must have completed a minimum of 11 of 14 nocturnal heartburn ratings during the run-in period (i.e. <=3 "missing" nocturnal heartburn ratings during the 14-day period)
* Patients must have a total nocturnal heartburn symptom score of >4 points during the 2-week run-in period
* 3 "missing" nocturnal heartburn ratings during the 14-day period) as recorded in the diary
* Night-time heartburn control assessment of "very dissatisfied, dissatisfied, neither dissatisfied nor satisfied" at the end of the 2-week run-in period.

Exclusion Criteria:

* Patients currently taking rabeprazole 20mg once daily (morning or evening administration) or 10mg twice daily (morning and evening administration) on a continuous basis
* Documented evidence of GERD refractory to acid suppressive therapy (i.e.
* no or poor clinical response to at least two treatment courses of 4-weeks duration with a PPI)
* Esophagitis known to be the result of systemic events (e.g. scleroderma, ingested irritants)
* Active GI bleeding, or presence of "alarm symptoms" (i.e., vomiting, blood in stool, anemia, dysphagia)
* Documented history of significant pyloric stenosis or esophageal ring stricture
* Documented evidence of esophageal or gastric varices
* Patients with primary motility disorders, infectious or inflammatory conditions of the small or large intestine, malabsorption syndromes, GI obstruction, history of gastrointestinal malignancy, definitive acid-lowering surgery or other esophageal, gastric or intestinal surgery (including vagotomy) except for simple closure of perforation
* Patients who are unable or unwilling to discontinue the use of prostaglandins (e.g. misoprostol), sucralfate, prokinetic agents (e.g. metoclopramide), anticholinergics, cholinergic agents or spasmolytics. Use of opiates may be continued if started at least 2 weeks before study admission and the dosage is consistent (± 25% for total opioid daily dose) throughout the study
* Treatment with high-dose systemic corticosteroids (>10mg/day prednisone equivalent) and NSAIDs, including COX-2 selective inhibitors, cannot be initiated at anytime during the study. However, patients taking corticosteroids and NSAIDs (including ASA) before study entry may continue these medications during the study, however, they must have been taking a stable dose (e.g. for oral medication, a consistent daily dose ± 25%) for at least 2 weeks before study admission and the dosage must be kept constant throughout the study. Occasional, intermittent use of NSAIDs for acute, self-limiting conditions (e.g. headache relief) is acceptable during the study
* >3 daytime episodes during any 7 consecutive days of the run-in period
* >1 severe or very severe daytime episode (i.e., more than 1 daytime heartburn episode rated >=3) during any 7 consecutive days of the run-in period
* Maximum total daytime heartburn score >5 during any 7 consecutive days of the run-in period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-07; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The primary analysis will be based on the mean nocturnal heartburn score observed after four weeks of drug administration for each of the three dosing regimens of rabeprazole.

SECONDARY OUTCOMES:
Nocturnal heartburn score at end of treatment/ 8 weeks; HRQoL and productivity outcomes 4 & 8 wks; rescue meds usage & compliance with study meds over entire study; day-time heartburn score 4 & 8 wks.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada

REFERENCES:
- See also: A randomized, controlled, parallel-group, open-label study to evaluate different dosing regimens of rabeprazole in controlling nocturnal heartburn symptoms in patients with gastroesophageal reflux disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=360&filename=CR005692_CSR.pdf